CLINICAL TRIAL: NCT00161460
Title: Colorectal Cancer Screening Intervention in UWPN Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Cynthia Ko, Associate Professor, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 26840-J; 1R21CA107157 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Neoplasia
Keywords: Colorectal cancer; Mass screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Study nurse contacts subjects who enroll in the intervention to provide detailed education about screening tests, to assess their risk for colorectal cancer, and to facilitate screening.
  Interventions: Behavioral: colorectal cancer screening intervention
- 2 (No Intervention): Patients who do not enroll receive usual care from their primary care providers.

INTERVENTIONS:
Behavioral: colorectal cancer screening intervention — Enrolled subjects receive tailored education from a registered nurse who also facilitates ordering and completion of screening tests
  Arms: 1

SUMMARY:
The purpose of this study is to determine if a prototype colorectal cancer screening program with the services of a cancer prevention specialist will increase utilization of appropriate colorectal cancer screening tests.

DETAILED DESCRIPTION:
Colorectal cancer is the second leading cause of cancer death in the United States. Colorectal cancer screening is widely recommended, but generally under-utilized. Previous studies have shown that only a minority of people over the age of 50 are screened for colorectal cancer with either fecal occult blood testing or flexible sigmoidoscopy. Barriers to screening include patient and provider-related factors. An innovative program to support primary care providers in providing necessary education about colorectal cancer screening, to provide reminders when screening tests are due, and to facilitate requesting and follow-up of screening tests may help address some of these barriers to providing screening services.

In this proposal, we will develop and implement a primary care based-colorectal cancer screening program to supplement clinical services provided in a primary care practice network. This network uses an electronic medical record and has established referral patterns for gastrointestinal endoscopy services, radiology, and pathology. In the proposed screening program, we will develop a colorectal cancer screening module to supplement the existing electronic medical record. This module will enable providers to review risk factors for colorectal cancer, prior screening history, and need for future screening in one easily accessible location. The information provided by this module will be supplemented by the services of a cancer prevention specialist. This person will oversee enrollment of patients into the program, provide patient education about colorectal cancer screening, and facilitate ordering or referral for screening or follow-up tests.

Outcome measures will include utilization of screening rates, patient knowledge about screening tests, and provider acceptance of the program. If successful, this program may be useful to other large primary care practices, and may also help to improve utilization of other types of cancer prevention services.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and over, enrolled for medical care in the UWPN clinics

Exclusion Criteria:

* Primary care physicians feel they would not benefit from colorectal cancer screening, unwilling or unable to complete study procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer screening test utilization | 6 months

SECONDARY OUTCOMES:
Knowledge about colorectal cancer screening tests | 2 months
Cancer worry score | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ko, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States